CLINICAL TRIAL: NCT02362776
Title: Metabolic Changes as a Diagnostic Indicator for Cancer
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Algemeen Ziekenhuis Vesalius (Other); Ziekenhuis Maas en Kempen (Other); Mariaziekenhuis Noord-Limburg (Other)
Responsible Party: Principal Investigator, Prof. dr. Michiel Thomeer, prof. dr., Hasselt University
Other Study IDs: 09/046U
Record Dates: First submitted 2013-12-10; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer; Lung Cancer
Keywords: NMR spectroscopy; metabolic changes; blood plasma; biomarker; cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Metabolic phenotype of cancer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- breast cancer patients
  Interventions: Other: Venous blood sample
- lung cancer patients
  Interventions: Other: Venous blood sample
- control subjects
  Interventions: Other: Venous blood sample

INTERVENTIONS:
Other: Venous blood sample — Collection of a venous blood sample to investigate metabolic changes in blood

SUMMARY:
This study aims to determine whether metabolic changes occur in blood plasma of cancer patients, and whether these changes can be used as a biomarker to detect cancer. These analyses will be done by means of nuclear magnetic resonance (NMR) spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast or lung cancer (new lesion)

Exclusion Criteria:

* Not fasted for at least 6 hours
* Plasma glucose concentration ≥ 200 mg/dl
* Intake of medication at the day of investigation
* History/treatment of cancer in the previous 5 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of breast or lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Metabolic phenotype of cancer | day 1
  Significant metabolic changes in blood between cancer patients & control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Thomeer, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg; Kurt Baeten, dr., Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Hasselt University, Hasselt, Limburg

REFERENCES:
- [Derived] Louis E, Adriaensens P, Guedens W, Vanhove K, Vandeurzen K, Darquennes K, Vansteenkiste J, Dooms C, de Jonge E, Thomeer M, Mesotten L. Metabolic phenotyping of human blood plasma: a powerful tool to discriminate between cancer types? Ann Oncol. 2016 Jan;27(1):178-84. doi: 10.1093/annonc/mdv499. Epub 2015 Oct 20. PMID 26487580